CLINICAL TRIAL: NCT04631783
Title: Is the Daytime Sleepiness Based on Epworth Sleepiness Scale a Good Way to Assess Taiwanese With Suspected Obstructive Sleep Apnea.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-09-006CC
Record Dates: First submitted 2020-11-15; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational survey with retrospective follow-up is designed to study the daytime sleepiness based on Epworth Sleepiness Scale a good way or not to assess Taiwanese with suspected obstructive sleep apnea.

DETAILED DESCRIPTION:
Daytime sleepiness (DS) is a complicated clinical problem, often indicating a serious underlying physiological abnormality and associated with higher prevalence of comorbid conditions such as diabetes, myocardial infarction, and stroke. Daytime sleepiness is also the cardinal symptoms of obstructive sleep apnea. How to identify the high risks patients with obstructive sleep apnea for further polysomnography is a difficult problem for doctors in out-patient department. Different methods have been proposed for measuring sleepiness and the Epworth sleepiness scale (ESS) is the measure of sleepiness most commonly used in sleep research and clinical settings.

However, whether Epworth sleepiness scale is a good tool with high predictive value of obstructive sleep apnea is not evaluated in the population of Taiwanese. This observational study is set up to document these practices.

ELIGIBILITY:
Inclusion Criteria:

* patients with polysomnography during 2016/1/1-2019/12/31

Exclusion Criteria:

* age under 20 year-old
* incomplete polysomnography
* incomplete chart information
* patients with narcolepsy
* patients with previous diagnosed with obstructive sleep apnea, including already patients with obstructive sleep apnea under treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with polysomnography during 2016/1/1-2019/12/31
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between Epworth sleepiness scale and the severity of obstructive sleep apnea | baseline (The Epworth sleepiness scale was completed just before the polysomnography)
  use analysis to calculate the correlation
The specificity and sensitivity of Epworth sleepiness scale for obstructive sleep apnea | Baseline (The Epworth sleepiness scale was completed just before the polysomnography)
  use receiver operating characteristic curve (cut point of 10) to calculate the specificity and sensitivity

SECONDARY OUTCOMES:
Questionnaire: If there are some specific symptoms as a tool with better sensitivity or specificity than Epworth sleepiness scale for obstructive sleep apnea | Baseline